CLINICAL TRIAL: NCT07366138
Title: Ultrasound-Guided External Oblique Intercostal Plane Block Versus Subcostal Transversus Abdominis Plane Block For Perioperative Analgesia in Laparoscopic Sleeve Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Alaa El din Ali, Resident of Anesthesiology, Egypt., Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS.28.12.2025
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Ultrasound; External Oblique Intercostal Plane Block; Subcostal Transversus Abdominis Plane Block; Perioperative Analgesia; Laparoscopic Sleeve Gastrectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EOIP Group (Group A ) (Experimental): Patients will receive an ultrasound-guided bilateral external oblique intercostal plane (EOIP) block using 20 mL of 0.25% bupivacaine in each side after induction of anesthesia and prior to surgical incision.
  Interventions: Other: External oblique intercostal plane block
- Subcostal TAP Group (Group T) (Experimental): Patients will receive a bilateral subcostal transversus abdominis plane (TAP) block using 20 mL of 0.25% bupivacaine in each side, under ultrasound guidance and identical conditions.
  Interventions: Other: Subcostal transversus abdominis plane block

INTERVENTIONS:
Other: External oblique intercostal plane block — Patients will receive an ultrasound-guided bilateral external oblique intercostal plane (EOIP) block using 20 mL of 0.25% bupivacaine in each side after induction of anesthesia and prior to surgical incision.
  Arms: EOIP Group (Group A )
Other: Subcostal transversus abdominis plane block — Patients will receive a bilateral subcostal transversus abdominis plane (TAP) block using 20 mL of 0.25% bupivacaine in each side, under ultrasound guidance and identical conditions.
  Arms: Subcostal TAP Group (Group T)

SUMMARY:
This study aims to compare the analgesic efficacy, duration of analgesia, and overall opioid consumption between the external oblique intercostal plane (EOIP) block and subcostal transversus abdominis plane (TAP) block in patients undergoing laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
Postoperative pain management is a critical aspect of enhanced recovery after surgery (ERAS) protocols, particularly in laparoscopic bariatric procedures such as sleeve gastrectomy.

Among the ultrasound-guided abdominal wall blocks, the transversus abdominis plane (TAP) block and its subcostal variant have demonstrated efficacy for upper abdominal surgeries. The subcostal TAP block provides analgesia for the T6-T9 dermatomes, covering incisions in upper abdominal procedures like laparoscopic cholecystectomy and bariatric surgery.

The external oblique intercostal plane (EOIP) block is a relatively new fascial plane block that targets the intercostal nerves lying between the external oblique and intercostal muscles.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both genders.
* American Society of Anesthesiologists (ASA) class I or II
* Body mass index (BMI) between 30-50 kg/m².
* Scheduled for elective laparoscopic sleeve gastrectomy under general anesthesia.
* Written informed consent from patients or surrogate decision makers.

Exclusion Criteria:

* Patient refusal.
* Allergy to local anesthetics.
* Coagulation disorders or anticoagulant therapy.
* Local infection or scar at the injection site.
* Severe hepatic or renal dysfunction.
* Chronic opioid use or psychiatric illness interfering with pain assessment.
* Conversion to open surgery or intraoperative complications requiring re-exploration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Patient-controlled analgesia (PCA) using intravenous morphine (1 mg bolus, 10-minute lockout) will be available for rescue analgesia when visual analogue score ( VAS ) > 3.

SECONDARY OUTCOMES:
Time to first rescue analgesia | 24 hours postoperatively
  Time to first rescue analgesia will be recorded from the end of surgery till first dose of morphine administrated.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the visual analogue score (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable").
  VAS will be recorded at 0, 2, 6, 12, and 24 hours postoperatively (at rest and cough).
Heart rate | Till the end of surgery (Up to two hours)
  Heart rate will be recorded intraoperatively and postoperatively
Mean arterial blood pressure | Till the end of surgery (Up to two hours)
  Mean arterial blood pressure will be recorded intraoperatively and postoperatively
Incidence of postoperative nausea and vomiting | 24 hours postoperatively
  Incidence of postoperative nausea and vomiting (PONV) will be recorded.
Block-related complications | 24 hours postoperatively
  Block-related complications such as pleural puncture, local anesthetic toxicity, and hematoma will be recorded.
Degree of patient satisfaction | 24 hours postoperatively
  Patient satisfaction will be assessed using a 5-point Likert scale at 24 hours (1 = very dissatisfied , 2 = dissatisfied, 3 =mild, 4= moderate satisfaction, 5 = very satisfied ).

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, Benha, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.